CLINICAL TRIAL: NCT06649500
Title: Comparison Between Treatment with Sensorized Treadmill and Conventional Therapy in Balance Disorders and Use of Artificial Intelligence in Identifying Predictive and Prognostic Indices of the Risk of Falling in Balance Disorders in Adult-elderly Subjects
Brief Title: Identify the Most Effective Rehabilitation Method Between a Treatment with a Sensorized Treadmill (Walker View) and a Treatment with Conventional Group Therapy in Balance Disorders and the Use of Artificial Intelligence to Identify Predictive Indices to Prevent Falls and Diagnose Promptly the Risk
Acronym: UAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Federica Bressi, Professor, Fondazione Policlinico Universitario Campus Bio-Medico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180.24 CET2cbm; PNC0000007 (Other Grant/Funding Number: Italian Ministry of Research, complementary actions NRRP "Fit4MedRob-Fit For Medicial Robotics")
Record Dates: First submitted 2024-10-14; First posted 2024-10-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Balance Disorders; Rehabilitation; Falls; Falls Prevention; Artificial Intelligence (AI); Elderly (people Aged 65 or More)
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Sensorized Treadmill (Experimental): Patients will carry out treatment with a sensorized treadmill, Walker View. This treadmill gives the possibility to patients to see their image reconstructed in a 3D mode in order to observe the bad aligments that increase the patients balance disorders. The feedback systems are necessary to give continuous stimulation to the patients.
  Each patients will carry out 18 treatment sessions and each session will last 30 minutes
  Interventions: Other: Treadmill
- Conventional Therapy (Active Comparator): Patients in this arm will carry out treatment with a conventional group therapy, consisting in usual treatment according to current clinical practice.
  Each patient will undergo 18 sessions of conventional therapy based on group re-education.
  Interventions: Other: conventional therapy
- Clinical monitoring (No Intervention): Patients in this arm will take part in the 'no intervention' part of the study and they will not carry out treatment. Patients will undergo only a clinical monitoring with an educational intervention, which does not elvove treatment or exercises, and they will continue to follow their daily habits.

INTERVENTIONS:
Other: Treadmill — The Walker View system is a treadmill equipped with a loaded cell sensor belt and a 3D camera that allows you to detect every single angular movement of the subject. Furthermore, thanks to the two optics, a classic one for 2D shooting in high resolution, and a revolutionary one for infrared rays, it is possible to reconstruct the position of the subject in space in three-dimensional mode and in real time. The reflected image reconstructed by the system helps to improve movement through the "continuous feedback system" method.
  Arms: Experimental Sensorized Treadmill
Other: conventional therapy — Conventional therapy intervention will follow the usual treatment according to current clinical practice. This treatment will be delivered to patients in a group session in order the balance disorders.
  Arms: Conventional Therapy

SUMMARY:
Falls in the elderly are one of the main sources of disability and hospitalization, with a significant impact on quality of life and social and healthcare costs. Falls represent a significant health concern for people over 60 years old. Numerous studies have shown that falls cause serious health consequences. Around 30% of people over the age of 60 experience a fall during the year.

According to the impact falls have, the investigators decided to analyze the effectiveness of training on a Walker View sensorized treadmill, with the possibility of exercises for coordination and balance, compared to training with a conventional group therapy, in order to understand the best training to reduce the risk of falling and observe the possible improvements in daily life activities.

So the study aims to identify the most effective rehabilitation method between a treatment with a sensorized treadmill (Walker View) and a conventional group therapy in balance disorders.

The study also aims to identify predictive indices, with the use of Artificial Intelligence, that can contribute to the prevention and diagnosis of balance disorders in a short time and prevent falls in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Consent to participate in the study
* Positive history of balance disorders
* Absence of cognitive deficits (MMSE ≥ 24)
* Tinetti < 25

Exclusion Criteria:

* Clinical pictures associated with musculoskeletal, cardiovascular, cerebrovascular, neuro-psychic problems and post-surgical outcomes that make the planned evaluation tests unfeasible.
* Inability to carry out a walking test.
* History of more than one fall in the last six months.
* Subjects who have not expressed informed consent to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Step Length of Gait Analysis | Baseline, 6 weeks, 10 weeks
  The Gait Analysis is used to assess individuals with conditions that affect their ability to walk. It is a useful test for studying gait, thanks to instruments that measure the load on each limb and walking in general. It allows us to evaluate progresses at different time frames.

SECONDARY OUTCOMES:
Balance | Baseline, 6 weeks, 10 weeks
  Balance will be assessed through the Tinetti Scale, a validated tool to measure balance skills, including risk of falls and walking in elderly subjects.
  Each item is given a score ranging from 0 to 2, where zero equals inability, 1 ability with aid or adaptation and 2 complete ability. A lower score indicates lower capabilities. A score < or equal to 18 indicates high risk of falling, 19-24 indicates medium risk of falling, > or equal to 25 low risk of falling.
Mobility | Baseline, 6 weeks, 10 weeks
  Mobility is assessed through the Time Up and Go Test that measures the level of mobility and requires static and dynamic balancing skills to perform the test
Risk of falling | Baseline, 6 weeks, 10 weeks
  Risk of falling is assessed through the Berg Scale used to assess balance and the risk of falling. 14 items will be evaluated, each item assigns a score from 0 to 4 (with 0 = unable to perform the task, 4 = able to perform the task within the times and conditions indicated). Scores below 20 points indicate the need for the patient to use a wheelchair or aids; scores between 21 and 45 suggest using an aid when walking; scores above 45 suggest patients are able to move safely without the need of aids.
Daily Living | Baseline, 6 weeks, 10 weeks
  Daily Living is assessed with the Barthel Index for Activities of Daily Living. It is an ordinal scale which measures a persons ability to complete activities of daily living (ADL) and it assesses functional independence. The scale assigns one point for each independent function in order to obtain a total performance result that varies from 0 (complete dependence) to 6 (independence in all functions).
Instrumental Activites of Daily Living | Baseline, 6 weeks, 10 weeks
  These activities will be assessed through the IADL scale and it respectively investigates the ability of elderly subjects to carry out fundamental functions of daily life. One point will be assigned for each independent function in order to obtain a total performance result that varies from 0 (complete dependence) to 8 (independence in all functions)
Muscle strength | Baseline, 6 weeks, 10 weeks
  This will be assessed with the Motricity Index which aims to measure muscle strength and motor skills at the limb level.
Patient reported Quality of Life | Baseline, 6 weeks, 10 weeks
  This will be assessed by the QoL scale SF-36. It measures 36 items in order to objectify to quantify health status and measure health-related quality of life. The aggregate scores for each domain range from 0 to 100, as a percentage, where the higher the score, the more favorable the health status.
Stability | Baseline, 6 weeks, 10 weeks
  This outcome measure will be assessed with the stabilometric platform, which measures the average position of the body's centre of gravity and its small movements around that position.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Campus Bio Medico di Roma, Rome, Rome, Italy